CLINICAL TRIAL: NCT01619683
Title: A 12 Month, Single Blind, Placebo Controlled, Phase III Study to Assess the Effects of Enclomiphene Citrate Treatment On Bone Mineral Density in Men With Secondary Hypogonadism
Brief Title: Assessment of the Effects of Enclomiphene Citrate on Bone Mineral Density in Men With Secondary Hypogonadism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single
Other Study IDs: ZA-303
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Effect of Treatment on Bone Mineral Density
MeSH Terms: interventions — Enclomiphene

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Androxal (Experimental)
  Interventions: Drug: enclomiphene citrate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: enclomiphene citrate — 12.5 mg, 1 capsule, daily, oral. After 6 weeks of treatment, subjects will remain on 12.5 mg/day if their morning testosterone level is greater than 300 ng/dL. If a subject's testosterone is less than 300 ng/dL, the subject's dose will be increased to 25 mg/day
  Other Names: Androxal
  Arms: Androxal
Drug: Placebo — 1 placebo capsule per day, oral
  Arms: Placebo

SUMMARY:
To determine the effects of 12 months of treatment with Androxal on bone mineral density in men with secondary hypogonadism.

DETAILED DESCRIPTION:
This study is a phase III single-blind placebo-controlled safety study with a 52 week active dosing period with Androxal. Safety will be assessed by physical and visual acuity exams, slit lamp and fundoscopy eye exams, clinical laboratory tests, DEXA scanning, lean soft tissue assessment (LST), and adverse event reporting. Results will be compared to an age-matched placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Overweight (BMI 25 to 42 kg/m2 inclusive, or BMI 23 to 42 inclusive in Asian subjects) males age 18 to 60 inclusive
2. Men currently using topical testosterone products should wash-out for at least 7 days before Visit 1
3. All clinical laboratory tests within normal ranges (any clinically significant deviation of laboratory results will require approval of sponsor)
4. Previously or concurrently diagnosed as having secondary hypogonadism and confirmed with morning testosterone <300ng/dL measured twice on separate days. One of the two TT levels must be confirmed at baseline. Subjects who fail this criterion will be enrolled in the placebo group.
5. LH <9.4 mIU/mL (at Visit 1 only)
6. Ability to complete the study in compliance with the protocol
7. Ability to understand and provide written informed consent

Exclusion Criteria:

1. Use of an injectable or pelleted testosterone within 6 months prior to study (men currently on topical products may be enrolled in the study after a 7-day washout period)
2. Use of testosterone injection, spironolactone, cimetidine, Clomid, 5α-reductase inhibitors, hCG, androgen, estrogen, anabolic steroid, DHEA, or herbal hormone products during the study
3. Use of Clomid in the past year
4. Uncontrolled hypertension or diabetes mellitus based on the Investigator's assessment at baseline. Subjects treated for Type II diabetes will be allowed into the study. Newly diagnosed diabetics need to be treated for at least 48 hours before being enrolled in the study
5. Clinically significant abnormal findings at screening (Visit 1), based on the Investigator's assessment.
6. A hematocrit >54% or a hemoglobin >17 g/dL
7. Clinically significant abnormal laboratory findings at baseline (Visit 2), based on the Investigator's assessment
8. Use of an investigational drug or product, or participation in a drug or medical device research study within 30 days prior to receiving study medication.
9. Known hypersensitivity to Clomid
10. Symptomatic cataracts (nuclear sclerosis cataract or cortical cataract grade > 2 based on 0-4 scale or any trace of posterior subcapsular cataract)
11. Abnormal fundoscopy exam such as central retinal vein occlusion
12. Any condition which in the opinion of the investigator would interfere with the participant's ability to provide informed consent, comply with study instructions, possibly confound interpretation of study results, or endanger the participant if he took part in the study
13. Irreversibly infertile or compromised fertility (cryptorchism, Kallman Syndrome, primary hypogonadism, or tumors of the pituitary)
14. Current or history of breast cancer
15. Subjects with a Z-score of <2
16. Hyperparathyroidism, metabolic bone disease, previous fracture of the spine, recent chemotherapy, use of medications that may influence BMD (thyroid replacement therapy, immunosuppressive therapy, prednisone or antiepileptic drugs
17. No intravenous or oral contrast agents within 7 days.
18. Subject weighs >300 pounds (>136 kg)
19. Current or history of prostate cancer or a suspicion of prostate disease unless ruled out by prostate biopsy, or a PSA>3.6
20. Presence or history of known hyperprolactinemia with or without a tumor
21. Chronic use of medications use such as glucocorticoids
22. History of drug abuse or chronic narcotic use including methadone
23. Subjects with known history of HIV and/or Hepatitis C
24. Subjects with end stage renal disease
25. Subjects with cystic fibrosis (mutation of the CFTR gene)
26. Enrollment in a previous Androxal study

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | 52 weeks
  Change in bome mineral density at the end of study compared to placebo

SECONDARY OUTCOMES:
Testosterone | 52 weeks
  Changes of values from baseline in total morning Testosterone levels at week 52.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tempe, Arizona
  - Mission Viejo, California
  - Newport Beach, California
  - Rancho Cucamonga, California
  - Clearwater, Florida
  - Fort Lauderdale, Florida
  - Jupiter, Florida
  - Miami, Florida
  - Miami Gardens, Florida
  - Henderson, Nevada
  - Lawrenceville, New Jersey
  - New York, New York
  - Rochester, New York
  - Houston, Texas
  - Salt Lake City, Utah

REFERENCES:
- See also: Sponsor's corporate web page — http://www.reprosrx.com